CLINICAL TRIAL: NCT05477979
Title: Cohort Studies of Associations of Psychological Stress With Therapy Efficacy and Prognosis of Lung Cancer, Including Non-small-cell Lung Cancer and Small-cell Lung Cancer With Early and Advanced Staging (STRESS-LUNG)
Brief Title: The Associations of Psychological Stress With Therapy Efficacy and Prognosis of Lung Cancer (STRESS-LUNG)
Status: Recruiting | Type: Observational
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Fang Wu, Professor, Central South University
Other Study IDs: XYEYY20220704
Record Dates: First submitted 2022-07-23; First posted 2022-07-28 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancer; Psychological Stress; Immune Checkpoint Inhibitors; Cancer, Treatment-Related
Keywords: Lung cancer; Immune checkpoint inhibitors; Psychological stress; Cancer progression; Prognosis; Biomarker
MeSH Terms: conditions — Lung Neoplasms; Stress, Psychological; Neoplasms, Second Primary; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1: advanced NSCLC patients receiving first-line ICIs (STRESS-LUNG-1 study): For stage IIIB-IV patients with NSCLC who have received immune checkpoint inhibitors as first-line therapy.
  Interventions: Other: Exposure: psychological stress status
- Cohort 2: limited-stage and extensive-stage SCLC patients receiving ICIs (STRESS-LUNG-2 study): For limited-stage and extensive-stage SCLC patients who have received immune checkpoint inhibitors
  Interventions: Other: Exposure: psychological stress status
- Cohort 3: NSCLC patients receive neoadjuvant therapy of ICIs（STRESS-LUNG-3 study）: For stage IB-IIIB patients with non-small cell lung cancer who have received neoadjuvant therapy of immune checkpoint inhibitors.
  Interventions: Other: Exposure: psychological stress status
- Cohort 4: NSCLC patients receive radical resection (STRESS-LUNG-4 study)): For early-stage patients with non-small cell lung cancer who have received radical resection.
  Interventions: Other: Exposure: psychological stress status

INTERVENTIONS:
Other: Exposure: psychological stress status — The assessment of depressive and anxiety symptoms was conducted using Patient Health Questionnaire-9 (PHQ-9) and Generalized Anxiety Disorder Assessment 7 (GAD-7). Patients with a PHQ-9 score ≥ 5 or a GAD-7 score ≥ 5 were categorized as the stressed group.

SUMMARY:
This is the prospective, observational cohort study (STRESS-LUNG) to explore the associations of psychological stress with progression, efficacy of immune checkpoint inhibitors (ICIs) and prognosis of Lung Cancer. The participants including the patients diagnosed with advanced non-small-cell lung cancer (NSCLC) who received the first-line therapy or neoadjuvant therapy of ICIs; patients diagnosed with advanced small-cell lung cancer (SCLC) receiving the first-line therapy ICIs; patients diagnosed with early small-cell lung cancer (SCLC) receiving surgery.

DETAILED DESCRIPTION:
This is the prospective, observational cohort study (STRESS-LUNG) to explore the associations of psychological stress with progression, efficacy of ICIs and prognosis of Lung Cancer. This study will have 4 cohorts

* Cohort 1 (STRESS-LUNG-1): A prospective, observational cohort study to explore the association between psychological stress and the efficacy of first-line treatment of ICIs in advanced NSCLC.
* Cohort 2 (STRESS-LUNG-2): A prospective, observational cohort study to explore the association between psychological stress and the efficacy of first-line treatment of limited-stage and extensive-stage SCLC.
* Cohort 3 (STRESS-LUNG-3): A prospective, observational cohort study to explore the association between psychological stress and the efficacy of neoadjuvant therapy of ICIs in resectable NSCLC.
* Cohort 4 (STRESS-LUNG-4): A prospective, observational cohort study to explore the association of psychological stress with cancer progression, and Prognosis in early-stage NSCLC receiving radical surgery.

ELIGIBILITY:
Cohort 1 (STRESS-LUNG-1):

Inclusion Criteria:

1. Age ≥ 18 years;
2. Histologically confirmed diagnosis of NSCLC;
3. Unresectable locally advanced, metastatic, or recurrent stage ⅢB-Ⅳ based on AJCC TNM staging 8th edition;
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
5. Systematic treatments naive ( e. g., chemotherapy, anti-angiogenic drugs, targeted drugs, and immunotherapy );
6. Presence of at least one measurable lesion according to the Response Evaluation Criteria in Advanced Solid Tumors version 1.1 (RECIST v1.1) ;
7. Receiving PD-1/PD-L1 inhibitors monotherapy or combination with chemotherapy;
8. Informed and agreed to participate in the study;

Exclusion Criteria:

1. Epidermal growth factor receptor (EGFR)-sensitizing mutation and/or anaplastic lymphoma kinase (ALK) gene and/or ROS proto-oncogene 1 (ROS1) fusion-positive;
2. Combined with other malignant tumors in the past 3 years;
3. Concurrent acute or chronic psychiatric disorders;
4. Current receiving anti-depressive or anti-anxiety therapy;
5. Previous treatment with other clinical drug trials;
6. Patients with symptomatic brain metastasis;
7. Can't cooperate with psychological scale assessment;

Cohort 2 (STRESS-LUNG-2):

1. Age ≥ 18 years；
2. Pathologically diagnosed as small cell lung cancer；
3. Unresectable locally advanced, metastatic, or recurrent stage Ⅲ-Ⅳ based on AJCC TNM staging 8th edition;
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
5. Systematic treatments naive ( e. g., chemotherapy, anti-angiogenic drugs, targeted drugs, and immunotherapy );
6. Presence of at least one measurable lesion according to the Response Evaluation Criteria in Advanced Solid Tumors version 1.1 (RECIST v1.1) ;
7. Receiving PD-1/PD-L1 inhibitors monotherapy or combination with chemotherapy;
8. Informed and agreed to participate in the study;

Exclusion Criteria:

1. Combined with other malignant tumors in the past 3 years;
2. Concurrent acute or chronic psychiatric disorders;
3. Current receiving anti-depressive or anti-anxiety therapy;
4. Previous treatment with other clinical drug trials;
5. Patients with symptomatic brain metastasis;
6. Can't cooperate with psychological scale assessment;

Cohort 3 (STRESS-LUNG-3):

1. Age ≥18 years ；
2. Pathologically diagnosed as non-small cell lung cancer;
3. Resectable clinical stage IB-IIIB based on AJCC TNM staging 8th edition;
4. At least one measurable lesion can be evaluated according to the RECIST 1.1 standard；
5. Systematic treatments naive ( e. g., chemotherapy, anti-angiogenic drugs, targeted drugs, and immunotherapy );
6. Receiving PD-1/PD-L1 inhibitors combined with chemotherapy as neoadjuvant therapy.

6. Cardiopulmonary function can withstand surgery; 7. Informed and agreed to participate in the study;

Exclusion Criteria:

1. Epidermal growth factor receptor (EGFR)-sensitizing mutation and/or anaplastic lymphoma kinase (ALK) gene and/or ROS proto-oncogene 1 (ROS1) fusion-positive;
2. Combined with other malignant tumors in the past 3 years;
3. Concurrent acute or chronic psychiatric disorders;
4. Current receiving anti-depressive or anti-anxiety therapy;
5. Previous treatment with other clinical drug trials;
6. Can't cooperate with psychological scale assessment;

Cohort 4 (STRESS-LUNG-4):

1. Age ≥18 years;
2. Pathologically diagnosed as non-small-cell lung cancer；
3. Pathologically stage conformed as early stage of IA-IIIA
4. Available for tumor tissue samples；
5. Systematic treatments naive ( e. g., chemotherapy, anti-angiogenic drugs, targeted drugs, and immunotherapy );
6. Receiving radical surgery;
7. Informed and agreed to participate in the study;

Exclusion Criteria:

1. Combined with other malignant tumors in the past 3 years;
2. Concurrent acute or chronic psychiatric disorders;
3. Current receiving anti-depressive or anti-anxiety therapy;
4. Previous treatment with other clinical drug trials;
5. Can't cooperate with psychological scale assessment;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants including the patients diagnosed with advanced non-small-cell lung cancer (NSCLC) who received the first-line therapy or neoadjuvant therapy of ICIs; patients diagnosed with advanced small-cell lung cancer (SCLC) receiving the first-line therapy ICIs; patients diagnosed with early small-cell lung cancer (SCLC) receiving surgery.
Sampling Method: Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Cohort 1 & 2: Progression-free survival (PFS) | 3 years
  Time from the beginning of first-line immunotherapy to the first progression (PD) in patients with lung cancer
Cohort 3: Pathologic complete response (pCR) rate | 3 years
  pCR is no viable tumor cells in tumor bed and lymph nodes. The pCR rate is the proportion of patients with a pathologic complete response.
Cohort 4: Disease-free survival (DFS) | 5 years
  The duration between the date after surgery to the date of any recurrence or death firstly

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  Overall survival (OS) is defined as the duration from the beginning of first-line immunotherapy until death due to any cause. Subjects who are still alive at the end of the study observation period will be censored at the time of last known vital status.
Quality of life | 5 years
  Quality of life (QoL) is assessed longitude by Short Form Health Survey 36 (SF-36) and EORTC QLQ-C30 (version.3).
  SF-36 includes 36 items and assesses the functional status and well-being on eight multi-item subscales. The total score on each SF-36 subscale ranges between 0 and 100. A greater score indicates better QoL.
  The EORTC QLQ-C30 is composed of 9 multi-item scales: 5 functioning scales (physical, role, cognitive, emotional, and social), a global QOL scale, and 3 symptom scales (fatigue, pain, and nausea/vomiting). All scales and single items are linearly transformed to an 0-100 scale. A higher score represents a better level of functioning.
Objective Response Rate (ORR) | 2 years
  The proportion of patients with a complete response or partial response to treatment according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1)

OTHER OUTCOMES:
The correlation between gut microbiota and chronic stress and the efficacy of ICIs | 5 years
  The baseline fetal is collected and assessed by 16S rRNA sequencing. And explore the association between gut microbiota and chronic stress and the efficacy of ICIs during the enrolled observation process.
The correlation between tumor microenvironment signature and chronic stress and the efficacy of ICIs | 5 years
  The baseline paraffin-embedded tissue is collected and assessed by multiplex immunohistochemistry, including T lymphocytes, B lymphocytes, NK lymphocytes, macrophagocyte, and DC cells. And explore the association between tumor microenvironment signature and chronic stress and the efficacy of ICIs during the enrolled observation process.
The correlation between peripheral stress biomarker and immune cells signature and chronic stress and the efficacy of ICIs | 5 years
  The baseline peripheral venous blood is collected. The stress biomarkers including epinephrine, norepinephrine, cortisol and ACTH. The peripheral immune cells signature and assessed by flow cytometry, including T lymphocytes, B lymphocytes, NK lymphocytes, macrophagocyte, and DC cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology, The Second Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zeng Y, Hu CH, Li YZ, Zhou JS, Wang SX, Liu MD, Qiu ZH, Deng C, Ma F, Xia CF, Liang F, Peng YR, Liang AX, Shi SH, Yao SJ, Liu JQ, Xiao WJ, Lin XQ, Tian XY, Zhang YZ, Tian ZY, Zou JA, Li YS, Xiao CY, Xu T, Zhang XJ, Wang XP, Liu XL, Wu F. Association between pretreatment emotional distress and immune checkpoint inhibitor response in non-small-cell lung cancer. Nat Med. 2024 Jun;30(6):1680-1688. doi: 10.1038/s41591-024-02929-4. Epub 2024 May 13. PMID 38740994